CLINICAL TRIAL: NCT04773743
Title: Feasibility of a Remotely Delivered Yoga Intervention for Chronic Low Back Pain
Brief Title: Remotely Delivered Yoga Program for Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maryland University of Integrative Health (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07.SUL.10.20.2
Record Dates: First submitted 2021-01-22; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain
Keywords: chronic pain; yoga; meditation
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronic nonspecific low back pain (Experimental): Remotely delivered yoga intervention
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Remotely delivered yoga intervention

SUMMARY:
The purpose of this research is to integrate the meditative components of integrative restoration (iRest) yoga nidra with simple and safe movement sequences derived from established yoga postures and physical therapy interventions for chronic nonspecific low back pain and to use telemedicine technology to facilitate the intervention in a diverse socioeconomic and racial/ethnic population. This project will first systematically adapt the iRest yoga intervention for the incorporation of movement using a consultative and iterative process followed by a pilot intervention to assess the acceptability and preliminary efficacy of this program for pain, back related function and to address body-mind regulation and biopsychosocial-spiritual well-being. Hypothesis: a yoga intervention emphasizing meditative movement and relaxation will be safe for remote delivery and effective for biopsychosocial-spiritual outcomes for people with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-64 years who report chronic nonspecific low back pain, defined as low back pain of unknown etiology persisting for at least 12 weeks,

  * Participants must report an average pain intensity in the previous week of 4 or greater on an 11-point (0 to 10) numerical rating scale,
  * Demonstrate medium to high risk on the STarT back screening tool,
  * Understand English
  * Have access to technology including a computer and internet access

Exclusion Criteria:

* Specific causes of low back pain (e.g. spinal fractures, cancer-related pain)

  * Severe or progressive neurological deficits
  * Severe chronic medical and/or psychiatric comorbidities that may prevent safe participation in the study
  * Established pregnancy
  * Current yoga practice or regular yoga class attendance in the last three months;
  * Current application for a receipt of workers compensation
  * lack of access to technology including a computer and the internet

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index | Pre, midpoint (4 weeks), final (8 weeks), 1 month follow up
  Back related function and pain

SECONDARY OUTCOMES:
Change in Vagal Efficiency | Pre, midpoint (4 weeks), final (8 weeks), 1 month follow up
  A device will be used to measure Heart rate variability and vagal efficiency
Change in Purpose in Life | Pre, midpoint (4 weeks), final (8 weeks), 1 month follow up
  Six item measure of purpose in life
Change in Body Brain Center Sensory Scales | Pre, midpoint (4 weeks), final (8 weeks), 1 month follow up
  Subjective measure of sensory sensitivity
Change in Body Perception Questionnaire subscale on autonomic reactivity | Pre, midpoint (4 weeks), final (8 weeks), 1 month follow up
  Subjective measure of autonomic reactivity

CONTACTS AND LOCATIONS:
Overall Officials: Marlysa Sullivan, MPT, Principal Investigator — Maryland University of Integrative Health

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data